CLINICAL TRIAL: NCT02178111
Title: Not Performing Episiotomy Versus Selective Episiotomy: a Randomized Clinical Trial
Brief Title: Comparison of Never Performing Episiotomy to Performing it in a Selective Manor
Acronym: EPISIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, MD PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPISIO
Record Dates: First submitted 2014-06-16; First posted 2014-06-30 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Need of Episiotomy
Keywords: episiotomy, vaginal delivery, randomized, perineum
MeSH Terms: interventions — Episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Never perform episiotomy (Experimental): In this group the birth attendant will sought to avoid the use of episiotomy, and try not to carry out the procedure unless considered absolutely needed
  Interventions: Other: Never perform episiotomy
- Selective episiotomy (Active Comparator): Patients will be subjected to the usual routine (selective episiotomy, ie, in the presence of indications described in the literature, according to the discretion of the physician or nurse assisting the birth)
  Interventions: Procedure: episiotomy

INTERVENTIONS:
Other: Never perform episiotomy — In this group birth attendants will be sought to avoid at all cost episiotomy. The intention is to never perform episiotomy in this group.
  Arms: Never perform episiotomy
Procedure: episiotomy
  Arms: Selective episiotomy

SUMMARY:
The study hypothesis is that not performing never episiotomies is safe and results are equivalent to performing episiotomies ina selective manor.

DETAILED DESCRIPTION:
World Health Organization recommends that the rate of episiotomy in various departments will be around 10%, which is already a reality in many European countries. The episiotomy should be limited and physicians should be encouraged to use their clinical judgment to decide when the procedure is necessary. There are no clinical evidence corroborating any indication of episiotomy, so not yet known whether episiotomy is indeed necessary in any context obstetric practice. Objectives: To compare the maternal and perinatal outcomes in women undergoing a protocol of not conducting episiotomy versus selective episiotomy. Methods: A randomized clinical trial will be conducted in open Maternity Instituto de Medicina Integral Prof. Fernando Figueira, from August 2012 to July 2013. 340 women will be included in labor with term pregnancy, maximum dilation of 8 cm, live fetus in cephalic vertex presentation and will be excluded women with bleeding disorders of pregnancy , indication for caesarean section, women without capacity to consent and without legal guardians. The primary outcomes will be: frequency of episiotomy, delivery duration, frequency of spontaneous lacerations, frequency of instrumental delivery. frequency of perineal trauma, postpartum blood loss, need for perineal suturing, number of sutures, Apgar scores at one and five minutes, need for neonatal resuscitation and pH in cord blood. As secondary outcomes will be assessed: frequency of severe perineal trauma, complications of perineal suturing perineal pain postpartum evaluated according to the visual scale, maternal satisfaction, neonatal morbidity and admission RN in NICU. Women will be invited to participate and those who agree should signing the consent form. At the beginning of the second stage will open the envelope to determine which group included women, with 170 assigned to a protocol of not conducting episiotomy (experimental group) and 170 to a group that episiotomy is performed selectively (Control Group ), according to the judgment of the provider of care delivery. Statistical analysis will be performed using the Epi-Info statistical program 7, adopting the principle of intention to treat. The analysis will be performed with the groups identified as A or B by a blinded statistician to the meaning of the lyrics, breaking the secrecy only after the results obtained and prepared the tables. Categorical variables were compared in contingency tables, using the chi-square test of association and Fisher's exact test, as appropriate. The risk ratio (RR) shall be calculated as measure of relative risk, determining the confidence interval at 95%. Regarding the quantitative variables, if they have normal distribution, comparison between groups will be conducted through the Student's t test for unpaired samples. If it is found that the distribution is not normal, the nonparametric Mann-Whitney-will be used. Ethical aspects, the present study addresses the Resolution 196/96 of the National Health Council and will be submitted to the iMIP Research Ethics Committee, beginning only after your approval. All participants will be included only if they agree to voluntarily participate by signing the consent

ELIGIBILITY:
Inclusion Criteria:

* Women in active labor admitted to the maternity ward
* Term pregnancy (37-42 weeks gestation);
* Maximum Dilation 8cm;
* Live fetus in vertex position.

Exclusion Criteria:

* hemorrhagic syndromes of pregnancy (premature separation of the normally implanted placenta
* Women with an indication for cesarean section: cephalopelvic disproportion (DCP), non reassuring fetal heart rate, dystocia;
* Women without capacity to consent and without legal guardians.
* Women undergoing cesarean delivery (post-randomization exclusion)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
duration of the second stage of labor | From beginning of second stage of labor to delivery of the baby
  Time in minutes from beginning of second stage of labor until the delivery of the baby
frequency of episiotomy | From diagnosis of second stage of labor to delivery of the neonate
  Frequency of episiotomies in fact carried out
frequency of spontaneous lacerations | From randomizatyion to one hour after delivery
  Frequency of spontaneous lacerations verified immediatly after delivery (time frame from randomization until one hour after delivery)
blood loss at delivery | from delivery to one hour postpartum
  Volume of blood loss in mililiters, lost by the patient from the genital tract, from the moment of the delivery to one hour after delivery
perineal need of suturing | From delivery to one hour postpartum
  Perineal suturing carried out by the birth attendant
Apgar scores | From delivery to five minutes after delivery
  one and five minutes Apgar scores
need for neonatal resuscitation | From delivery to one hour after delivery
  Need of any resuscitation procedures carried out in the conduction of the neonate, from the time of birth until one hour after delivery
cord blood pH at birth | From birth of the baby until first minute after delivery
  Cord blood pH ( hydrogen ion concentration) at birth collected just after delivery

SECONDARY OUTCOMES:
frequency of severe perineal trauma | from delivery of the baby until one hour after delivery
  frequency of severe perineal trauma observed by the birth attendant
complications of perineal suture | From delivery until 15 days after delivery
  presence of hematoma, or infection or dehiscence of perineal suture described in the patients records from the moment of the delivery until 15 days after the delivery
perineal pain after childbirth | From 24 hours after delivery until 48 hours of the delivery
  perineal pain after childbirth evaluated according to the visual scale and maternal satisfaction, the evaluation is carried from 24 to 48 hours after the delivery, before maternal discharge from the hospital
admission of the newborn (NB) in the neonatal intensive care unit (ICU). | from delivery until 28 days after birth
  admission of the newborn (NB) in the neonatal intensive care unit (ICU).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Inês Melo, MS, Principal Investigator — IMIP
Locations (1):
- IMIP, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] M Amorim M, Coutinho IC, Melo I, Katz L. Selective episiotomy vs. implementation of a non-episiotomy protocol: a randomized clinical trial. Reprod Health. 2017 Apr 24;14(1):55. doi: 10.1186/s12978-017-0315-4. PMID 28438209
- [Derived] Melo I, Katz L, Coutinho I, Amorim MM. Selective episiotomy vs. implementation of a non episiotomy protocol: a randomized clinical trial. Reprod Health. 2014 Aug 14;11:66. doi: 10.1186/1742-4755-11-66. PMID 25124938